CLINICAL TRIAL: NCT00000392
Title: Phase II Study of the Efficacy of Peptide T in HIV-Positive Individuals With Cognitive Impairment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH00013
Record Dates: First submitted 2000-01-17; First posted 2000-01-18 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2013-10

CONDITIONS: HIV Infections; Cognition Disorders
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Cognition Disorders; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Peptide T

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Peptide T (Active Comparator): Peptide T given intranasally at a dosage of 2mg 3 times a day for 6 months
  Interventions: Drug: Peptide T
- Placebo (Placebo Comparator): Placebo given intranasally at a dosage of 2mg 3 times a day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Peptide T
  Arms: Peptide T
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the chemical efficacy and safety of intranasally administered peptide T on neurocognitive function in HIV seropositive individuals.

Previous studies have shown that treatment with peptide T can result in cognitive improvement in HIV-infected patients.

Patients are randomized to receive either peptide T or placebo for the first 6 months. All patients then receive open-label peptide T for approximately 6 additional months. Neuropsychologic tests are used to determine drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have:

  1. Cognitive dysfunction on neuropsychological testing.
  2. HIV antibody positivity.
  3. Expected survival of 6 months.
  4. EITHER no use of an antiretroviral within the past 4 weeks OR use of approved regimens of AZT, ddI, or ddC.
  5. Medically stable EKG and urinalysis.
  6. Given informed, written consent to participate.
* Allowed:

  1. Inhaled aerosolized pentamidine for Pneumocystis carinii pneumonia prophylaxis, dapsone, cotrimoxazole, topical antifungal agents, nystatin or ketoconazole, acyclovir.
  2. Amitriptyline (up to 50 mg/day) or an equivalent dose of another antidepressant for relief of peripheral neuropathy that is expected to remain unchanged throughout the first 6 months of the study.
* Abstinence or agree to use barrier methods of birth control / contraception during the study
* Negative pregnancy test within 30 days of study entry
* Bilirubin <= 3
* CD4 (Must be <= 500 cells/mm3 if patient is without non-cognitive HIV-related symptoms. CD4 count > 500 cells/mm3 allowed if patient has other (non-cognitive) HIV-related symptoms. ( 0 - 100 - 200 - 300 - 400 - 500 - 600 - 700 - 800 plus.)
* Creatinine <= 1.5 mg/dl
* Granulocytes >= 750
* Hemoglobin > 8 g/dl (No more than two transfusions per month permitted.)
* Other Lab Values Prothrombin time > 70 percent of control.
* Platelet Count >= 75000 /mm3
* SGOT(AST) < 5 x ULN (ULN = upper limit of normal).

Exclusion Criteria:

* Patients with the following are excluded:

  1. History of mental retardation or learning disability.
  2. Evidence of current DSM-III-R Axis I disorder within 3 months prior to study entry or past history of psychotic disorder or bipolar mania.
  3. History of neurologic disorder not secondary to HIV infection (e.g., head trauma requiring medical observation or hospitalization, seizure disorder).
* Patients with the following symptoms or conditions are excluded:

  1. Kaposi's sarcoma or other malignancy likely to require chemotherapy during the first 6 months of the study.
  2. Serious underlying medical problems that may complicate interpretation of the treatment results, including unstable diabetes mellitus, severe arteriosclerotic heart disease, uncontrolled hypertension, or hepatic or renal failure.
  3. Non-HIV related condition that is likely to interfere with interpretation of neuropsychologic test results.
  4. Inability to participate in neuropsychologic testing or unable to comply with intranasal study medication administration.
* Excluded within 4 weeks prior to study entry:

  1. Antiretrovirals except as allowed in the Patient Inclusion Criteria.
  2. Psychoactive agents (e.g., benzodiazepines, antidepressants, antipsychotics, amphetamines)

Excluded within 8 weeks prior to study entry:

Long-acting psychoactive agents (e.g., Prozac).

* Active alcohol abuse in the past 3 months, or abuse judged by the investigators as likely to interfere with the analyses of neuropsychologic function. Abuse of cocaine, marijuana, heroin or other opiates (including methadone), barbiturates, amphetamines or other substances within the past 3 months, judged by the investigators as likely to interfere with the analyses of neuropsychologic tests.
* Positive pregnancy test within 30 days of study entry
* No abstinence or no agreement to use barrier methods of birth control / contraception during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 1990-01; Primary Completion 1996-08 (Actual); Study Completion 1996-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCSD, San Diego, California
  - Univ of Miami School of Medicine, Miami, Florida

REFERENCES:
- [Background] Heseltine PN, Goodkin K, Atkinson JH, Vitiello B, Rochon J, Heaton RK, Eaton EM, Wilkie FL, Sobel E, Brown SJ, Feaster D, Schneider L, Goldschmidts WL, Stover ES. Randomized double-blind placebo-controlled trial of peptide T for HIV-associated cognitive impairment. Arch Neurol. 1998 Jan;55(1):41-51. doi: 10.1001/archneur.55.1.41. PMID 9443710

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 457 persons screened for cognitive impairment, 205 men and 10 women were randomized (106 to peptide T and 109 to placebo).
Groups:
- Peptide T: Peptide T given intranasally at a dosage of 2mg 3 times a day for 6 months
  Peptide T
- Placebo: Placebo given intranasally at a dosage of 2mg 3 times a day for 6 months
  Placebo
Period: Overall Study
Arm/Group | Peptide T | Placebo
Started | 106 | 109
Completed | 66 (provided complete NP outcome data constituted the sample for the primary efficacy analyses) | 77 (provided complete NP outcome data constituted the sample for the primary efficacy analyses)
Not Completed | 40 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peptide T | Placebo | Total
Number analyzed (Participants) | 106 | 109 | 215
Age, Customized [Number; unit: Participants] — Information is not available for all participants.
  Participants
    18-39 years | 60 | 62 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 101 | 104 | 205
Race/Ethnicity, Customized [Number; unit: Participants] — Information is not available for all participants.
  Participants
    White | 83 | 94 | 177
    Hispanic | 16 | 9 | 25
    Black | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 106 | 109 | 215

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Neurocognitive Performance z Score From Baseline
Description: Higher values for change in z-score represent an improvement in Neurocognitive Performance (NP)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: z score
Arm/Group | Peptide T | Placebo
Number analyzed (Participants) | 66 | 77
z score | 0.24 (0.05) | 0.16 (0.03)
Statistical Analysis 1: Comparison: Peptide T vs Placebo; Test type: Superiority or Other; p = 0.18, ANOVA

2. Secondary Outcome: Change in Neurocognitive Performance Domain z Scores From Baseline
Description: Higher values for change in z-score represent an improvement in Neurocognitive Performance (NP)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: z score
Arm/Group | Peptide T | Placebo
Number analyzed (Participants) | 66 | 77
z score
  Verbal fluency | 0.14 (0.09) | 0.15 (0.08)
  Visuospatial ability | 0.17 (0.06) | 0.25 (0.06)
  Abstract thinking | 0.34 (0.07) | 0.23 (0.04)
  Speed of information processing | 0.23 (0.07) | 0.14 (0.05)
  Working memory | 0.23 (0.09) | 0.08 (0.07)
  Learning and retention | 0.19 (0.07) | 0.11 (0.06)
  Motor performance | 0.19 (0.06) | 0.18 (0.06)

ADVERSE EVENTS:
Description: Only data for the events that were statistically significant between the two treatment groups could be retrieved because adverse event data are lost.
Arm/Group | Peptide T | Placebo
Serious Adverse Events (participants affected / at risk) | 8/106 | 3/109
Other Adverse Events (participants affected / at risk) | 75/106 | 57/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peptide T (N=106) | Placebo (N=109)
Death (Immune system disorders) | 8 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peptide T (N=106) | Placebo (N=109)
Depression or Irritability (Psychiatric disorders) | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 34 | 42
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Proteinuria (Renal and urinary disorders) | 18 | 9
Eosinophilia (Blood and lymphatic system disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No